CLINICAL TRIAL: NCT03347058
Title: Immunotherapy & Me
Acronym: IO & Me
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Support Community, Research and Training Institute, Philadelphia (Other)
Responsible Party: Principal Investigator, Heather Badt, MBA, President, Cancer Support Community, Cancer Support Community, Research and Training Institute, Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CSC-IO-0102
Record Dates: First submitted 2017-11-06; First posted 2017-11-20 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cancer
Keywords: immunotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive programming (Other): Access to a suite of resources, including digital tools, person-to-person support, and educational resources
  Interventions: Other: Supportive programming

INTERVENTIONS:
Other: Supportive programming — Access to a suite of resources, including digital tools, person-to-person support, and educational resources

SUMMARY:
Immunotherapy & Me is a pilot study to determine patient and provider needs around immunotherapy treatment, and to determine the most meaningful resources to improve patient outcomes and decrease cost. Specifically, this study aims:

1. To determine whether layering in customizable resources at the point-of-care that offer healthcare providers care-management tools to give their immunotherapy patients leads to changes in (a) patients' knowledge, attitudes, and health behaviors (including self-reported measures of self-efficacy and empowerment, cancer-related distress, quality of life, and satisfaction with the programs offered) and (b) improved clinical outcomes (including decreased hospital admissions, decreased hospital readmissions, and decreased costs associated with hospitalizations).
2. To successfully integrate the Immunotherapy & Me program within oncology practices to provide a model framework for dissemination across other care providers. Once success is demonstrated, a turn-key model of immunotherapy patient support can be expanded to other oncology care systems.

DETAILED DESCRIPTION:
As usage and indications for immunotherapy increase, there presents a critical need to identify patient-centered and practice solutions across the continuum of care. Immunotherapy & Me is an innovative program of customizable resources that seeks to improve the patient experience by supporting the unique needs of both immunotherapy patients and the clinical staff who care for them. The Cancer Support Community (CSC) will implement this operational framework of patient and provider tools at multiple geographically and demographically diverse oncology practices.

The program will include CancerSupportSource® (CSS), a self-administered screening instrument for individuals with cancer that takes approximately 10 minutes to complete and has been validated in 300 English-speaking cancer survivors at CSC affiliates nationwide.The instrument consists of cancer-related problems (physical, social, psychological, emotional and practical) and has been demonstrated to have good internal consistency reliability. Patients are asked to rate the severity of their concerns and if they would like to talk with a staff person and/or receive additional information about their concerns. This information is used to address immediate concerns as well as to develop ongoing educational experiences that are tailored and integrated with their care.

At the end of year one, CSC will evaluate program impact, retool interventions as necessary, and pursue additional funding with the goal of extending services at existing practice sites - and scaling this turnkey model of immunotherapy treatment support.

ELIGIBILITY:
Inclusion Criteria:

* Receiving immunotherapy as a cancer treatment at a participating pilot site location
* English- or Spanish-speaking, or having access to a translator

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
CancerSupportSource® | One year
  Cancer-related distress
# of ER visits | One year
  Measured via self-report through a questionnaire developed for this study issued every 30 days
# of hospitalizations | One year
  Measured via self-report through a questionnaire developed for this study issued every 30 days

SECONDARY OUTCOMES:
Self-reported patient confidence in accessing resources | One year
  Measured with a Likert scale (Not at all confident to Extremely confident); assessed every 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Linda House, RN, BSN, MSM, Principal Investigator — Cancer Support Community
Locations (5):
- United States (5):
  - Catholic Health Initiatives, Englewood, Colorado
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - OHC, Cincinnati, Ohio
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - West Cancer Center, Germantown, Tennessee

IPD SHARING:
Plan to Share IPD: No